CLINICAL TRIAL: NCT05997667
Title: A Prospective, Multicenter, Randomized Controlled Clinical Study Evaluating the Efficacy and Safety of Rechargeable Implantable Deep Brain Stimulation System for the Treatment of Parkinson's Disease
Brief Title: Study on the Efficacy and Safety of Rechargeable Implantable DBS System in the Treatment of Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lepu Medical Technology (Beijing) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LPDBS-2023
Record Dates: First submitted 2023-08-07; First posted 2023-08-18 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Parkinson Disease
Keywords: Rechargeable implantable deep brain stimulation (DBS) system; Parkinson's disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Subjects in this arm will receive stimulation of DBS system within 1 month after surgery.
  Interventions: Device: Rechargeable implantable deep brain stimulation system
- control group (Other): Subjects in this arm will receive stimulation of DBS system at 3 months after surgery.
  Interventions: Device: Rechargeable implantable deep brain stimulation system

INTERVENTIONS:
Device: Rechargeable implantable deep brain stimulation system — The DBS system will be implanted in subjects in both study arms. Subjects in experimental group will receive stimulation of DBS system within 1 month after surgery.
  Arms: experimental group
Device: Rechargeable implantable deep brain stimulation system — The DBS system will be implanted in subjects in both study arms. Subjects in control group will receive stimulation of DBS system at 3 months after surgery.
  Arms: control group

SUMMARY:
The purpose of this clinical trial is to verify the efficacy and safety of rechargeable implantable deep brain stimulation (DBS) system for the treatment of advanced primary Parkinson's disease.

DETAILED DESCRIPTION:
This study is a prospective, multicenter, randomized controlled superiority clinical study. According to the unified inclusion and exclusion criteria, 60 eligible subjects are enrolled in this clinical trial. All subjects are implanted with bilateral deep brain stimulation leads, and are randomly assigned to the experimental group or control group in a 1:1 ratio. Within one month after surgery, the DBS system of experimental group is activated and the stimulation parameters are modulated, whereas the control group is not activated. The primary endpoint is the change in motor examination scores evaluated using the Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) part III (MDS-UPDRS-III) in "med off" state at 3 months after surgery, compared to the baseline. After primary endpoint evaluation, both groups receive treatment with activated DBS system. The efficacy in med off/stim on and med on/stim on state and the safety are evaluated at 6 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 years old, male or female;.
2. Primary PD (according to the UK Parkinson's Disease Society Brain Bank clinical diagnostic criteria for primary PD or Chinese diagnostic criteria for primary PD), with a duration of PD ≥ 4 years, and the improvement rate after an acute levodopa challenge test ≥ 30%; or primary PD, mainly characterized by tremor, the improvement of tremor by standardized drug treatment is not satisfactory and tremor is severe, which affects the patients' quality of life, after evaluation, duration can be relaxed to 3 years, the improvement rate of acute levodopa challenge test can be<30%.
3. The use of levodopa once had good effects, but currently cannot satisfactorily control symptoms (significant decrease in efficacy or occurrence of fluctuations in motor function or motor dysfunction), which affects quality of life.
4. Good compliance, patients and their families have the willingness to participate in the clinical trial of "bilateral implantation surgery of nervous stimulation system", voluntarily participate in this trial and sign informed consent form, patients can follow up regularly, and can accurately complete of assessment items, or the family members, guardians, or caregivers may assist the patients.

Exclusion Criteria:

1. Severe cognitive impairment (MMSE score: illiterate<17, elementary school<20, junior high school or above<24), poor compliance due to dementia, and/or inability to sign informed consent form
2. Patients with a history of severe mental illness and a Hamilton Depression Scale (HAMD) score>24
3. Seizure history in the last 1 year
4. Patients with severe heart, liver and kidney diseases, severe hypertension and severe orthostatic hypotension that affect their health status.
5. Patients with severe diabetes or serious cardiovascular and cerebrovascular diseases that affect their health status
6. Confirmed malignant tumor
7. Patients with surgical contraindications (e.g., the presence of active implants (whether turned on or not), or the presence of non-active implants that may affect the deep brain stimulation system, stereotactic nucleus lesioning, etc.), or other surgical procedures within six months that the researchers believe have an impact on this trial, or other neurosurgery contraindications
8. Patients who have suffered a previous cranial neurological injury
9. Women who are pregnant or preparing for pregnancy
10. Patients with severe alcohol dependence and drug abuse
11. Patients who received electric shock therapy within 30 days before surgery
12. Patients who are abnormally sensitive to temperature or who are allergic to heat
13. Subjects who are currently participating in other clinical trials or have participated in other clinical studies that have not reached the primary endpoint within three months.
14. Patients who are not suitable to participate in this clinical study in the opinion of the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-07-20 (Actual); Primary Completion 2025-01-20 (Estimated); Study Completion 2025-07-20 (Estimated)

PRIMARY OUTCOMES:
Change in motor examination score evaluated using the Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part Ⅲ in "med off" state relative to baseline | 3 months after surgery
  MDS-UPDRS Part Ⅲ (MDS-UPDRS-Ⅲ) scores range from 0 to 132, higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Change in motor examination score evaluated using the Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part Ⅲ in "med on" state relative to baseline | 3 months after surgery
  MDS-UPDRS Part Ⅲ (MDS-UPDRS-Ⅲ) scores range from 0 to 132, higher scores mean a worse outcome.
Change in motor experiences of daily living score evaluated using the Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part Ⅱ relative to baseline | 3 and 6 months after surgery
  MDS-UPDRS Part Ⅱ (MDS-UPDRS-Ⅱ) scores range from 0 to 52, higher scores mean a worse outcome.
Change in non-motor experiences of daily living score evaluated using the Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part Ⅰ relative to baseline | 3 and 6 months after surgery
  MDS-UPDRS Part Ⅰ (MDS-UPDRS-Ⅰ) scores range from 0 to 52, higher scores mean a worse outcome.
Change in motor complications score evaluated using the Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part Ⅳ relative to baseline | 3 and 6 months after surgery
  MDS-UPDRS Part Ⅳ (MDS-UPDRS-Ⅳ) scores range from 0 to 24, higher scores mean a worse outcome.
Change in "ON" time and "OFF" time relative to the baseline | 3 and 6 months after surgery
Change in motor examination score evaluated using the Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part Ⅲ with stimulation in "med on" and "med off" states relative to baseline | 6 months after surgery
  MDS-UPDRS Part Ⅲ (MDS-UPDRS-Ⅲ) scores range from 0 to 132, higher scores mean a worse outcome.
Change in daily levodopa equivalent dose relative to baseline | 3 and 6 months after surgery
Change in the Parkinson's Disease Questionnaire (PDQ-39) score relative to baseline | 6 months after surgery
  The Parkinson's Disease Questionnaire (PDQ-39) is a 39-item questionnaire designed to measure the specific impact of PD on quality of life. Scores range from 0 to 156, higher scores mean a worse outcome.
Evaluation of equipment operational performance | Within surgery, 1 month and 3 months after surgery
  The operational performance of the equipment is evaluated as excellent, good, or poor.
Incidence of adverse events | up to 6 months after surgery

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - ZhuJiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - The Second Affiliated Hospital of Air Force Medical University, Xi'an, Shaanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang